CLINICAL TRIAL: NCT00001951
Title: Hormone Replacement in Young Women With Premature Ovarian Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000045; 00-CH-0045
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2006-10

CONDITIONS: Healthy; Osteoporosis; Premature Ovarian Failure
Keywords: Bone; Cognition; Estrogen; Mood; Testosterone; Osteoporosis; Ovarian Failure; Hormone Replacement Therapy; POF; Premature Ovarian Failure
MeSH Terms: conditions — Osteoporosis; Primary Ovarian Insufficiency

INTERVENTIONS:
Drug: TMTDS

SUMMARY:
The human ovary produces male sex hormones (androgen) and female sex hormones (estrogen). Currently, androgen is not included in hormone replacement therapy for women with premature ovarian failure. Present hormone replacement therapy (HRT) was designed to treat women who experience ovarian failure at menopause (around the age of 50). However, 1% of women will experience premature failure of the ovaries before the age of 40. There have been no studies conducted to determine proper hormone replacement therapies for these younger women. Some research suggests that the usual menopausal hormone replacement therapy is not adequate to protect young women with premature ovarian failure from developing osteoporosis. Women with premature ovarian failure have abnormally low levels of androgens circulating in their blood. This may contribute to the increase risk for osteoporosis.

This study will compare two treatment plans for women with premature ovarian failure. Treatment plan one will be physiological estrogen hormone replacement. Treatment plan two will be physiological estrogen hormone replacement plus androgen. The study will attempt to determine which plan is more beneficial to women in relation to osteoporosis and heart disease.

The hormones will be contained in patches and given by placing the patches against the patient's skin. The patches were designed to deliver the same amount of hormone as would be normally produced by the ovary in young women.

The success of the treatment will be measured by periodically checking the density of patient's bone in the leg (femoral neck bone) . Researchers will take an initial (baseline) measurement of bone density before beginning treatment and then once a year, for 3 additional years, during treatment. The study will also consider bone density of the spine, bone turnover, heart disease risk factors, and psychological state.

DETAILED DESCRIPTION:
Present menopausal hormone replacement therapy regimens were designed for women who experience ovarian failure around age 50. At least 1% of women, however, experience premature ovarian failure before the age of 40, but there have been no studies establishing optimal hormone replacement therapy regimens for these younger women. Available evidence suggests that the usual menopausal hormone replacement therapy is not adequate to protect young women with premature ovarian failure from developing osteoporosis. Women with premature ovarian failure have abnormally low circulating androgen levels, which may contribute to their risk for osteoporosis. We plan to compare physiological estrogen replacement with physiological estrogen plus androgen replacement in young women with premature ovarian failure to determine which regimen is more beneficial for bone mineral density and other metabolic parameters related to the risk for cardiovascular disease. This study employs transdermal estradiol and testosterone "patches" designed to deliver the same amount for each sex steroid normally produced by the ovary in young women in a physiological manner. Women with premature ovarian failure will be randomized to receive either estradiol plus placebo patches or estradiol plus testosterone patches. Both groups will receive cyclic progestin treatment. A group of age-matched women with normal ovarian function will serve as contemporaneous controls for bone density and other study measures. The primary outcome parameter is femoral neck bone mineral density, to be assessed at baseline, and after 1, 2, and 3 years of treatment. Other outcome parameters include lumbar spine bone mineral density, markers of bone turnover, cardiovascular disease risk factors, and cognitive function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with karyotypically normal spontaneous premature ovarian failure (as defined by screening protocol 91-CH-0127, i.e. women who have at least 4 months of amenorrhea, two FSH levels above 40 mIU/ml, at least one month apart, and a normal 46, XX karotype, diagnosed with premature ovarian failure prior to the age of 40) who are between the age of 18 and 42 years will be candidates.

EXCLUSION CRITERIA:

General:

Smokers (more than 2 cigarettes per day).

Alcohol users (more than 2 drinks of alcohol per day).

Body mass index (BMI, kg/m(2)) greater than or equal to 30 and less than or equal to 19.

Previous history of hip fracture or other active hip pathology.

Abnormalities of the hip precluding the assessment of bone mineral density.

Major dermatologic disorders, or a history of skin sensitivity to adhesive bandages, tape or transdermal matrix patches.

Hirsutism score greater than 8.

Acne score greater than 1.

Hysterectomy

Baseline free testosterone (FT) levels above the normal range (greater than 6.3 pg/ml in our current essay) and/or SHBG levels less than 36 nmol/L.

Medical use:

Any prior treatment in the past 6 months known to affect bone other than estrogen (i.e., calcitonin, biphosphonates, fluoride, anabolic steroids, testosterone, or herbal therapy that contains androstenedione, and DHEA).

Current and/or past use of: diuretics, anticoagulants (heparin, Coumadin), glucocorticoid drugs, gonadotropin-releasing hormone agonist or antagonist therapy, chemotherapy.

Medical history of:

Anorexia nervosa, hyperprolactinemia, insulin-dependent diabetes, Cushing's syndrome, gastrectomy, osteogenesis imperfecta, mastocytosis, rheumatoid arthritis, long-term parenteral nutrition, hemolytic anemia, hemochromatosis and thalassemia, ankylosing spondylitis, multiple myeloma, Vitamin D deficiency, Paget's disease, primary hyperparathyroidism, hyperthyroidism, hypothyroidism, any cancer or any other major illness.

Contraindications to hormone replacement therapy:

Thromboembolic event associated with previous estrogen use History of endometrial cancer or hyperplasia

History of breast cancer

Hypertriglyceridemia (fasting triglyceride levels greater than 500 mg/dL)

LDL greater than 190mg/dl

Patients taking "statins"

Serum Alkaline phosphatase greater than or equal to 2X the upper limit of normal

Serum GGT greather than or equal to 2X the upper limit of normal

Abnormal values on two or more hepatic panel tests

Undiagnosed Vaginal Bleeding

Known sensitivity to agents

Note: We will include patients with premature ovarian failure on antidepressant medications, since today's most common antidepressant medication (Prozac) does not have a major import on cognitive function. However, we will note whether they are on these medications.

CONTROL SELECTION CRITERIA:

Healthy non-pregnant regularly menstruating women (cycles between 21 and 35 days), non-smokers, non-alcohol users, under no medications, using non-hormonal contraceptive methods (i.e. barrier methods of contraception, or sterilization) and with no intention to conceive within the following 3 years.

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250
Dates: Start 1999-12; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kalantaridou SN, Davis SR, Nelson LM. Premature ovarian failure. Endocrinol Metab Clin North Am. 1998 Dec;27(4):989-1006. doi: 10.1016/s0889-8529(05)70051-7. PMID 9922918
- [Derived] Popat VB, Calis KA, Kalantaridou SN, Vanderhoof VH, Koziol D, Troendle JF, Reynolds JC, Nelson LM. Bone mineral density in young women with primary ovarian insufficiency: results of a three-year randomized controlled trial of physiological transdermal estradiol and testosterone replacement. J Clin Endocrinol Metab. 2014 Sep;99(9):3418-26. doi: 10.1210/jc.2013-4145. Epub 2014 Jun 6. PMID 24905063
- [Derived] Guerrieri GM, Martinez PE, Klug SP, Haq NA, Vanderhoof VH, Koziol DE, Popat VB, Kalantaridou SN, Calis KA, Rubinow DR, Schmidt PJ, Nelson LM. Effects of physiologic testosterone therapy on quality of life, self-esteem, and mood in women with primary ovarian insufficiency. Menopause. 2014 Sep;21(9):952-61. doi: 10.1097/GME.0000000000000195. PMID 24473536